CLINICAL TRIAL: NCT01141127
Title: Tranexamic Acid (TXA) During Pediatric Cardiac Surgery: A Prospective Randomised Study Comparing Two Dosing Regimens
Brief Title: Tranexamic Acid (TXA) in Pediatric Cardiac Surgery
Acronym: Exacyl
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CCML-2010-01; 2010-018301-11 (EudraCT Number)
Record Dates: First submitted 2010-06-04; First posted 2010-06-10 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Bleeding
Keywords: tranexamic acid in pediatric surgery; fibrinolysis and paediatric cardiac surgery
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- INTERMITENT ADMINISTRATION (Active Comparator): Administration of 10 mg/kg of Tranexamic Acid at the beginning ,the middle and at the end of the intervention
  Interventions: Drug: Tranexamic Acid
- continuous administration of Tranexamic Acid (Experimental): Administration of 10 mg /Kg of Tranexamic Acid at the beginning in the priming pump and continuous infusion of 1 mg/KG of Tranexamic Acid until the end of the intervention
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — Comparison of two dosage regimen of Tranexamic Acid

SUMMARY:
The purpose of this study is to determine tranexamic acid plasma levels in children undergoing cardiac surgery at risk of bleeding and to compare two dosing regimens.

DETAILED DESCRIPTION:
Tranexamic acid (TXA) is administered intravenously to prevent bleeding associated with cardiac surgery and by pass in adult and children. The pharmacokinetic of this product is unknown in the pediatric population. Only a few studies report a clinical efficacy with different dosages. The purpose of this study is to determine the plasma level of TXA using two different administrations methods: continuous versus intermittent. The second objective is to determine whether fibrinolysis decreased. The population consists in children weighting 10 to 30 Kilos, undergoing cardiac surgery and at high risk of bleeding.

ELIGIBILITY:
Inclusion Criteria:

* children weighing between 10 and 30kg surgery with cardiopulmonary bypass for congenital heart disease deemed hemorrhagic

Exclusion Criteria:

* the patients undergoing a surgical procedure short and simple
* patients with past history of convulsions neurologiques especially allergies to the TA
* patients with renal insufficiency

Ages: 12 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Preoperative plasma tranexamic acid concentration is measured using high performance liquid chromatography | Blood samples are collected during the operative period within 24 hours

SECONDARY OUTCOMES:
preoperative plasma tranexamic acid concentration is measured using high performance liquid chromatography | blood samples collected during the operative period within the first 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Roland COUTURIER, MD, Principal Investigator — CCML
Locations (1):
- Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson, France

REFERENCES:
- [Derived] Couturier R, Rubatti M, Credico C, Louvain-Quintard V, Anerkian V, Doubine S, Vasse M, Grassin-Delyle S. Continuous or discontinuous tranexamic acid effectively inhibits fibrinolysis in children undergoing cardiac surgery with cardiopulmonary bypass. Blood Coagul Fibrinolysis. 2014 Apr;25(3):259-65. doi: 10.1097/MBC.0000000000000051. PMID 24418941